CLINICAL TRIAL: NCT05337345
Title: A Phase I, Open-Label, Randomized, Two-part Parallel Study to Compare the Pharmacokinetics of Single Subcutaneous Injections of Cendakimab Administered Using Autoinjector Versus Using Prefilled Syringe, and to Evaluate the Pharmacokinetics of Cendakimab When Administered by Autoinjector at Different Injection Sites, in Healthy Participants
Brief Title: A Study to Evaluate the Drug Levels of Cendakimab Delivered Subcutaneously in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM042-003
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Cendakimab
MeSH Terms: interventions — cendakimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental)
  Interventions: Drug: Cendakimab
- Part 2 (Experimental)
  Interventions: Drug: Cendakimab

INTERVENTIONS:
Drug: Cendakimab — Specified Dose on Specified Days
  Other Names: CC-93538; BMS-986355; RPC4046

SUMMARY:
The purpose of this study is to evaluate the drug levels of cendakimab delivered subcutaneously in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants as determined by no clinically significant deviation from normal in medical history, physical examination, vital signs, ECGs, and clinical laboratory determinations
* Body Mass Index (BMI) of 18.0 to 30.0 kg/m2, inclusive. BMI = weight (kg)/[height (m)]2
* Body weight ≥40.0 kg

Exclusion Criteria:

* History of clinically significant infection within 4 weeks of dosing on Day 1
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory determinations beyond what is consistent with the target population
* History of clinically significant allergic reaction to any drug, biologic, food or vaccine

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to Day 105
Area under the concentration-time curve (AUC) from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to Day 105
AUC from time zero extrapolated to infinite time (AUC(INF)) | Up to Day 105

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) | Up to Day 107
Number of Participants with Adverse Events (AEs) | Up to Day 107
Number of participants with clinical laboratory abnormalities | Up to Day 107
Number of participants with vital sign abnormalities | Up to Day 107
Number of participants with physical examination abnormalities | Up to Day 107
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 107
Number of participants with concomitant medications | Up to Day 107
Number of participants with concomitant procedures | Up to Day 107
Time of maximum observed concentration (Tmax) | Up to Day 105
Terminal half-life (T-HALF) | Up to Day 105
Apparent total body clearance (CL/F) | Up to Day 105

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Anaheim Clinical Trials Llc, Anaheim, California, United States

REFERENCES:
- [Derived] Zhang P, De Oliveira CHMC, Yu K, Basdeo S, Charriez CM, Syto M, Thomas M, Murthy B. Pharmacokinetic Characterization of Cendakimab Administered with Different Devices and at Different Injection Sites in Healthy Participants. Eur J Drug Metab Pharmacokinet. 2025 Jul;50(4):307-317. doi: 10.1007/s13318-025-00949-0. Epub 2025 May 15. PMID 40374841
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm